CLINICAL TRIAL: NCT02186314
Title: Effect of Right Bifocal Ventricular Cardiac Pacing on Serum Level Natriuretic Peptides in Patients With Heart Failure and Pacemaker Indication
Brief Title: Effect of Right Bifocal Ventricular Cardiac Pacing on Serum Level Natriuretic Peptides in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Carolina Crhistianini Mizzaci, Effect of right bifocal cardiac ventricular pacing on serum level natriuretic peptides in patients with heart failure and pacemaker indication, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 4381
Record Dates: First submitted 2014-06-16; First posted 2014-07-10 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Heart Failure
Keywords: atrial fibrillation, heart failure, pacemaker
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apical stimulation (Active Comparator): Pacemaker Biotronik: apical stimulation
  Interventions: Device: Pacemaker Biotronik: apical stimulation; Device: Pacemaker Biotronik: bifocal stimulation
- Bifocal stimulation (Active Comparator): Pacemaker Biotronik: bifocal stimulation
  Interventions: Device: Pacemaker Biotronik: apical stimulation; Device: Pacemaker Biotronik: bifocal stimulation

INTERVENTIONS:
Device: Pacemaker Biotronik: apical stimulation — Patients with pacemaker (Biotronik): an electrode will be implanted in the apical position of the right ventricle and an electrode implanted in the septal position of the right ventricle.The patients will remained in apical stimulation for two months, after that they will be subjected to evaluation. At the end of the evaluation, patients will undergo cross-over groups( bifocal stimulation) and patients will be kept in the new pacing mode for two months when they will be submitted to clinical, laboratory evaluation and assessment of pacemaker
Device: Pacemaker Biotronik: bifocal stimulation — Patients with pacemaker (Biotronik): an electrode will be implanted in the apical position of the right ventricle and an electrode implanted in the septal position of the right ventricle.The patients will remained in bifocal stimulation for two months, after that they will be subjected to evaluation. At the end of the evaluation, patients will undergo cross-over groups( apical stimulation) and patients will be kept in the new pacing mode for two months, when they will be submitted to clinical, laboratory evaluation and assessment of pacemaker

SUMMARY:
In this study we will select twenty patients with chronic atrial fibrillation and ventricular dysfunction with permanent cardiac pacemaker indication. We will dosage serum level natriuretic peptides for comparison between conventional and bifocal cardiac pacing.

DETAILED DESCRIPTION:
The target study population will comprise patients with permanent atrial fibrillation with mild or moderate myocardial dysfunction according to the American consensus echocardiography and the classical indication for pacemaker by Brazilian Guidelines for Cardiac Implantable Electronic Devices Guidelines and the American Heart Association. Primary goal: Assess whether resynchronization achieved by bifocal right ventricle pacing has influence on serum levels of natriuretic peptides and whether this could be used as a measure of success. Secondary goal: To compare clinical parameters,compare electrocardiographic parameters (QRS complex stimulated) in ventricular apical position and ventricular bifocal position, assess quality of life by questionnaire Minnesota Living With Heart Failure. Will be implanted pacemaker endocardial bifocal, with placement of a ventricular endocardial electrode in the septal region and another in right ventricle apical, as adopted in the conduct of Pacemaker sector under local anesthesia and sedation. After pacemaker implantation, patients will be randomized in a 1:1 ratio to apical or bifocal stimulation. Patients remained in this mode of stimulation for two months, after which they will be subjected to the following sequence of reviews: Clinical assessment (functional classification of heart failure);assessment of quality of life by the Minnesota Living With Heart Failure Questionnaire, 12-lead electrocardiogram at rest, with measurements of stimulated QRS duration, evaluation of the parameters of the pacemaker, serum level of peptides. At the end of this period of evaluation, patients will undergo cross-over groups, those in apical ventricular pacing will be allocated in the bifocal group and the last one will be allocated to apical ventricular pace. Patients will be retained in the new pacing mode for two months, and at the end of this period will be submitted to clinical, laboratory and assessment of pacemaker evaluation as well. At the end of the study, all patients will be kept in bifocal ventricular pacing, as advocated in the conduct of Pacemaker sector.

ELIGIBILITY:
Inclusion Criteria:

* Permanent atrial fibrillation with bradycardia and classic indication for permanent pacemaker
* mild or moderate ventricular dysfunction (35% <left ventricle ejection fraction <55%) of any etiology
* Signature of the free and informed consent

Exclusion Criteria:

* Age <18 years
* left ventricle ejection fraction > 55% or ≤ 35%
* classic indication of cardiac resynchronization therapy by Brazilian Guidelines for Cardiac Implantable Electronic Devices
* Patients with left ventricle ejection fraction ≤ 35%, with permanent atrial fibrillation, heart failure with functional class III or IV despite optimal pharmacological treatment and QRS> 150 ms
* Patients with left ventricle ejection fraction ≤ 35%, with permanent atrial fibrillation, heart failure with functional class III or IV despite optimal pharmacological treatment and QRS 120-150 ms with evidence of dyssynchrony by imaging method
* Patients with indication for pacemaker when ventricular pacing is essential, left ventricle ejection fraction ≤ 35% and heart failure with functional class III or IV
* Refusal to signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Serum level of natriuretic peptides | 2 months
  Assess whether resynchronization achieved by bifocal right ventricle pacing has influence on serum levels of natriuretic peptides and whether this could be used as a marker of success.

SECONDARY OUTCOMES:
Clinical parameters | 2 months
  We will compare clinical parameters by New York Heart Association functional classification
Electrocardiographic parameters | 2 months
  We will compare electrocardiographic parameters (QRS complex stimulated) in ventricular apical position and ventricular bifocal position
Assess quality of life | 2 months
  We will evaluate quality of life: Minnesota Living with Heart Failure Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: carolina Mizzaci, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Carolina Christianini Mizzaci, São Paulo, São Paulo, Brazil